CLINICAL TRIAL: NCT03253588
Title: Clinical Outcome of Laparoscopic Tubal Preservation Surgery for Ectopic Pregnancy
Brief Title: Laparoscopic Tubal Preservation Surgery
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Stella Ting Wan Hua, Principal Investigator, Far Eastern Memorial Hospital
Other Study IDs: 106002-E
Record Dates: First submitted 2017-08-15; First posted 2017-08-18 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Ectopic Pregnancy
MeSH Terms: conditions — Pregnancy, Ectopic | interventions — Salpingostomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: laparoscopic salpingotomy or salpingostomy — A 3-port technique (2 x 5-mm and 1 x 10-mm trocars) was implemented. A diluted solution of vasopressin (20IU in 100 mL saline solution) was initially injected into the mesosalpinx of the affected tube, followed by a linear incision which allowed the removal of the gestational tissue. In case of a ruptured tubal pregnancy, the ectopic mass was evacuated directly from the ruptured site using a combination of forceps and suction device. The tubal lumen was either closed with a single-layer of continuous absorbable suture (salpingotomy) or left to heal by secondary intention (salpingostomy).

SUMMARY:
Traditionally, salpingectomy has been the standard procedure for managing ectopic pregnancy. We would like to evaluate the safety and efficacy of laparoscopic tubal preservation surgery in treating ectopic pregnancies (salpingostomy or salpingotomy) while preserving the fertility outcome of the patients, as well as to identify the factors predicting the presence of persistent ectopic pregnancy after the surgery.

DETAILED DESCRIPTION:
All surgically-treated ectopic pregnancies in women aged 20 and above between 01 January 2009 and 31 December 2016 were identified. Cases receiving laparoscopic salpingostomy or laparoscopic salpingotomy were extracted from the database, patient characteristics and surgical outcomes (changes of serumβ-hcg, presence of persistent ectopic pregnancy and subsequent management, subsequent pregnancy) were reviewed from their medical records. Univariate and multivariate logistic regression analysis were employed to predict the presence of persistent ectopic pregnancy after laparoscopic tubal preservation surgery.

ELIGIBILITY:
Inclusion Criteria:

* women who had laparoscopic tubal preservation surgery (including salpingostomy and salpingotomy) for ectopic pregnancy between January 2009 and November 2016

Exclusion Criteria:

* women with ectopic pregnancy at sites other than fallopian tube (i.e. interstitial, ovary, abdomen)

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women diagnosed with ectopic pregnancies and underwent laparoscopic tubal preservation surgery (including salpingostomy and salpingotomy)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
peri- and post-operative parameters | between January 2009 and November 2016
  success rate of tubal preservation surgery (defined by postoperative serum bcg <5 IU/mL), postoperative complications (number of women who had adverse surgical outcome such as bladder injury, bowel injury, massive bleeding), pregnancy outcome (number of women who conceived successfully following the intervention)

SECONDARY OUTCOMES:
factors affecting the surgical success rate | between January 2009 and November 2016
  relationship between patient's baseline characteristics and rate of persistent ectopic pregnancy (unvariate and multivariate analysis)

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Taipei, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No